CLINICAL TRIAL: NCT04180852
Title: Investigating Nutrition and Functional Outcome in Critically Ill Patients
Acronym: INFO
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Christian Stoppe, Principal Investigator, University Hospital, Aachen
Other Study IDs: 19-001
Record Dates: First submitted 2019-11-07; First posted 2019-11-29 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Neurosurgical Patients; Elderly Patients; Obese Patients; Cardiac Surgery Patients; Abdominal Surgery Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Neurosurgical patients: Non-elective admission to the neurosurgical ICU with one of the following acute intracranial pathologies which also serve as predefined subgroups:
  1. Intracranial hemorrhage (subarachnoid, subdural hemorrhage or intracerebral hemorrhage)
  2. Acute and severe head trauma with an initial Glasgow Coma Scale ≤10
  Interventions: Other: Functional tests without clinical consequence for the patients therapy
- Elderly patients: Age ≥ 70 years, predefined subgroups: ≥ 70 years and ≥80 years
  Interventions: Other: Functional tests without clinical consequence for the patients therapy
- Obese patients: BMI ≥ 35 kg/m2, furthermore predefined subgroups of patients with BMI ≥ 40 kg/m2 and BMI ≥ 45 kg/m2
  Interventions: Other: Functional tests without clinical consequence for the patients therapy
- Cardiac surgery patients: Admission to the cardiosurgical ICU after one of the following procedures using cardiopulmonary bypass, which also serve as predefined subgroups:
  1. Coronary revascularization (coronary artery bypass graft)
  2. Heart valve surgery
  3. Combined or complex heart surgery
  Interventions: Other: Functional tests without clinical consequence for the patients therapy
- Abdominal surgical patients: Admission to the abdominal surgery ICU after abdominal surgery
  Interventions: Other: Functional tests without clinical consequence for the patients therapy

INTERVENTIONS:
Other: Functional tests without clinical consequence for the patients therapy — Battery of tests, which measure the patients functional outcomes regarding their muscle mass, their muscle strength, fat mass, physical function, neuropsychological function and quality of life.

SUMMARY:
This is a single-center, multi-ICU prospective observational trial evaluating current nutritional practice and its influence of the physical function of critically ill patients.

DETAILED DESCRIPTION:
The investigators propose a prospective observational, single-center, multi-intensive care unit trial to evaluate the influence of current nutritional practice on the physical outcome in critically ill patients. At least 100 consecutive patients requiring surgery, who are admitted to any surgical ICU at the University Hospital RWTH Aachen will be recruited. Nutritional practices, such as dosage, timing and route of administration of the nutrition, as well as complications regarding the nutrition will be recorded and analyzed longitudinally from ICU-admission until hospital discharge. Patient outcomes, such as ICU- and hospital length of stay, duration of mechanical ventilation, organ dysfunction, complications and infections will be evaluated. To assess physical function of the patient, muscle mass, muscle strength, the ability of the patient to self-mobilize and perform every day activities will be measured.

This observational trial aims to assess the current standard of nutritional practice in the ICU, to detect problems and complications and to gather first evidences about the influence of nutrition on the physical function of the patient. This study also aims to compare the outcome of the predefined subgroups of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Adult patients (≥ 18 years)
* Patients admitted to a surgical ICU requiring surgical Intervention
* Patients requiring sedation and invasive ventilation for ≥ 48 hours
* Patients with an expected ICU-length of stay ≥ 72 hours

Exclusion Criteria:

* Pregnant or lactating patients
* Patients already receiving an intense nutrition support (home parenteral or enteral nutrition) in addition to normal nutrition on hospital admission
* Patients with disabling disease (neurological or physical) that prevents them from walking, sitting or standing before ICU admission
* Patients unable to follow orders from the study personnel (language barriers, neurological, psychiatric disorders)
* Death expected within 96 hours after admission due to severity of disease
* Enrolment in an industry sponsored randomized trial within the last 30 days (co-enrolment in academic randomized trials will be considered on a case by case basis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a clinical trial, which will include critically ill patients after informed consent. Patients who admitted to a surgical ICU following surgery or requiring surgery can be screened and included by our team. The general eligibility criteria are listed above. We will recruit patients, who can be classified as one of the following groups: a) neurosurgical Patients, b) elderly patients, c) obese patients, d) cardiac surgery patients and e) abdominal surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Nutritional status - basic demographics | at Study inclusion
  Chart review
Nutritional Status - nutritional screening | intensive care unit (ICU) admission, up to 1 week
  Nutritional Risk Screening 2002 (Score: 0-7; if ≥3 patient at nutritional risk)
Nutritional Status - nutritional risk in the critically ill (NUTRIC) | ICU admission, up to 1 week
  NUTRIC score (Score 0-10; if interleucin-6 (IL6) available 0-5=low malnutrition risk; if IL6 not available 0-4= at low malnutrition risk
Nutritional Status - Waist and mid-arm circumferences | Study inclusion, up to 1 week
  Waist and mid-arm circumferences
Differences of dosage of nutrition | until discharge from intensive care unit, an average of 30 days
  Cumulative delivery of macronutrients by infusion rates
Differences of dosage of nutrition | until discharge from intensive care unit, an average of 30 days
  Cumulative delivery of macronutrients by cumulative count of macronutrients
Differences of dosage of nutrition | until discharge from intensive care unit, an average of 30 days
  Cumulative delivery of macronutrients by nutrition used
Timing of nutrition | until discharge from intensive care unit, an average of 30 days
  Chart Review- start and stop times
Timing of nutrition - reason for discontinuation | at discharge from intensive care unit, an average of 30 days
  Chart review
Differences in route of administration of nutrition | discharge from intensive care unit, an average of 30 days
  Rates of oral, enteral and parenteral nutrition, feeding tubes and catheters used for nutrition
Incidence of Gastrointestinal symptoms | discharge from intensive care unit, an average of 30 days
  Chart review (vomiting, nausea, high gastric residual volumes, diarrhea, obstipation, aspiration, ileus, bowel ischemia)
Incidence Blood work irregularities | discharge from intensive care unit, an average of 30 days
  Chart review (electrolyte imbalance, blood sugar imbalance, dyslipidemia)
Incidence of Refeeding syndrome | discharge from intensive care unit, an average of 30 days
  Chart review
Incidence of complications related to the route of administration | discharge from intensive care unit, an average of 30 days
  Chart review (central venous catheter infection, misplaced and dislocated enteral feeding tubes)
Nutrition adequacy | discharge from intensive care unit, an average of 30 days
  Rates of energy and protein received in comparison to nutritional targets Chart review
Change in Muscle mass - Mid-arm circumference (MAC) | Study inclusion, discharge from intensive care unit and hospital discharge, up to 3 months
  MAC
Change in Muscle mass - Quadriceps thickness | Study inclusion, discharge from intensive care unit and hospital discharge, up to 3 months
  ultrasound
Change in Muscle mass - Quadriceps cross sectional area | Study inclusion, discharge from intensive care unit and hospital discharge, up to 3 months
  ultrasound
Change in Muscle strength - Handgrip strength | discharge from intensive care unit and hospital discharge, up to 3 months
  Dynamometry
Change in Muscle strength - Quadriceps strength | discharge from intensive care unit and hospital discharge, up to 3 months
  Dynamometry
Change in Physical function - Functional Status Score for the ICU | discharge from intensive care unit and hospital discharge, up to 3 months
  Functional Status Score for Intensive Care Unit (FSS-ICU) (Score 0-35; the higher the score, the better physical functioning)
Change in Physical function - Short Physical Performance Battery | discharge from intensive care unit and hospital discharge, up to 3 months
  Short Physical Performance Battery (SPPB) (Score: 0-12; 0=worst performance and 12=best performance)
Change in Physical function - 6-Minute Walk Test | discharge from intensive care unit and hospital discharge, up to 3 months
  6-minute walking distance
Change in Physical function - Manual Muscle Testing (MMT) | discharge from intensive care unit and hospital discharge, up to 3 months
  MMT
Change in Physical function - Katz Activities of Daily Living (ADL) | Hospital discharge, day 30 after study inclusion, up to 3 months
  ADL (Score: 0-100; the higher the more independent)
Change in Physical function - Lawton Instrumental Activities of Daily Living (IADL) | Hospital discharge, day 30 after study inclusion, up to 3 months
  IADL (score 0-8; the higher the more independent)
Change in Physical function - Clinical Frailty Score (CFS) | Study inclusion, Hospital discharge, day 30 after study inclusion, up to 3 months
  CFS (score 1-9; 1= Very fit and 9=terminally ill)
Change in Fat mass | Study inclusion, discharge from intensive care unit and hospital discharge, up to 3 months
  Thigh and abdominal fat (ultrasound)
Change in Neuro-psychological function - Mini Mental State Examination (MMSE) | discharge from intensive care unit, Hospital discharge, day 30 after study inclusion, up to 3 months
  MMSE (Score 0-30; 30= no dementia and <9= severe dementia)
Change in Neuro-psychological function - Becks Depression Inventory (BDI) | discharge from intensive care unit, Hospital discharge, day 30 after study inclusion, up to 3 months
  BDI (Score 0-63; 0= no depression and 63= severe depression)
Quality of life - Short Form 36 (SF-36) | day 30 after study inclusion
  SF-36 (Score: 0-100; 100=no limitation in daily life and 0=completely limited)
Quality of life - Living location | day 30 after study inclusion
  Rates of patients being discharged to nursing home, rehabilitation, home care etc. Discharge location used as surrogate for physical fitness after hospital discharge.

SECONDARY OUTCOMES:
Mortality Rate | up to 30 days after study inclusion
  Mortality
Length of stay - intensive care unit length of stay | discharge from intensive care unit, an average of 30 days
  ICU length of stay
Length of stay - Hospital length of stay | Hospital discharge, an average of 60 days
  Hospital length of stay
Readmission - ICU readmission rate | Hospital discharge, day 30 after study inclusion, up to 3 months
  ICU readmission rate
Readmission - Hospital readmission rate | up to 30 days after study inclusion, up to 3 months
  Hospital readmission rate
Change in acute organ dysfunction - sepsis-related organ failure assessment (SOFA score) | up to discharge from intensive care unit, an average of 30 days
  daily records (score 0-24; 0=normal function and 24= massively impaired function)
Acute organ dysfunction - hemodynamic parameters | up to discharge from intensive care unit, an average of 30 days
  blood pressure in mmHg
Acute organ dysfunction - hemodynamic parameters | up to discharge from intensive care unit, an average of 30 days
  vasopressors, cumulative dosage in ml/d
Acute organ dysfunction - hemodynamic parameters | up to discharge from intensive care unit, an average of 30 days
  heart rate bpm
Acute organ dysfunction - incidence of ventilation | up to discharge from intensive care unit, an average of 30 days
  mode of ventilation
Acute organ dysfunction - duration of ventilation | up to discharge from intensive care unit, an average of 30 days
  hours of ventilation
Acute organ dysfunction - sedation | up to discharge from intensive care unit, an average of 30 days
  duration of sedation in hours
Acute organ dysfunction - sedation | up to discharge from intensive care unit, an average of 30 days
  dosage of sedation, cumulative dosage in ml/d
Acute organ dysfunction - Richmond Agitation Scale | up to discharge from intensive care unit, an average of 30 days
  Richmond Agitation Scale (score: +4 - -5; +4=aggressive behavior, 0=calm,-5=not reacting to verbal or physical approaches)
Acute organ dysfunction - Confusion Assessment Method for the ICU (CAM-ICU) | up to discharge from intensive care unit, an average of 30 days
  CAM-ICU (score: 0-10; more than 2 errors= delirium)
Persistent Organ Dysfunction - Incidence of mechanical ventilation | Hospital discharge, day 30 after study inclusion, up to 3 months
  need for ventilation
Persistent Organ Dysfunction - Incidence of hemodynamic parameters | Hospital discharge, day 30 after study inclusion, up to 3 months
  vasopressors
Persistent Organ Dysfunction - Incidence of renal replacement therapy | Hospital discharge, day 30 after study inclusion, up to 3 months
  renal replacement therapy
Complications - Rate of surgical reevaluation | Hospital discharge, day 30 after study inclusion, up to 3 months
  surgical reevaluation
Complications - Rate of hemorrhage | Hospital discharge, day 30 after study inclusion, up to 3 months
  hemorrhage
Complications - Rate of thromboembolic events | Hospital discharge, day 30 after study inclusion, up to 3 months
  thromboembolic events
Complications - Rate of cardiovascular events | Hospital discharge, day 30 after study inclusion, up to 3 months
  cardiovascular events
Complications - Rate of infection | Hospital discharge, day 30 after study inclusion, up to 3 months
  infection
Complications - Rate of sepsis | Hospital discharge, day 30 after study inclusion, up to 3 months
  sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No